CLINICAL TRIAL: NCT00760617
Title: Observer-blind Safety and Immunogenicity Study of GlaxoSmithKline Biologicals' Influenza Vaccine GSK2186877A When Administered to Elderly Subjects.
Brief Title: Evaluation of Safety and Immunogenicity of GSK Biologicals' Influenza Vaccine GSK2186877A in Adults 65 Years and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 111737
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Results first posted 2012-04-23 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2016-10

CONDITIONS: Influenza
Keywords: Influenza; Elderly
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- New generation influenza vaccine GSK2186877A Group (Experimental): Subjects aged ≥65 years received 1 dose of New generation influenza vaccine GSK2186877A
  Interventions: Biological: GSK Bio's influenza vaccine GSK2186877A
- Fluarix elderly Group (Active Comparator): Subjects aged ≥65 years received 1 dose of Fluarix vaccine
  Interventions: Biological: Fluarix
- Fluarix young Group (Active Comparator): Subjects aged 18-40 years received 1 dose of Fluarix vaccine
  Interventions: Biological: Fluarix

INTERVENTIONS:
Biological: GSK Bio's influenza vaccine GSK2186877A — Intramuscular (IM) administration, 1 dose
  Arms: New generation influenza vaccine GSK2186877A Group
Biological: Fluarix — Intramuscular (IM) administration, 1 dose
  Arms: Fluarix elderly Group; Fluarix young Group

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of GlaxoSmithKline Biologicals' influenza vaccine GSK2186877A in adults 65 year of age and older.

This protocol posting deals with objectives & outcome measures of the extension phase at year 1. The objectives & outcome measures of the primary phase are presented in a separate protocol posting (NCT number = 00540592).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* A male or female aged 18-41 years or ≥65 years at the time of the vaccination and who participated in the 110847 study and completed the 6 month follow-up.
* Written informed consent obtained from the subject.
* Fee of acute aggravation of the health status as established by clinical evaluation (medical history and medical history directed examination) before entering into the study.
* Female subjects must be of non-childbearing potential.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days prior to vaccination, or planned use during the study period.
* Administration of other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrolment in this study. Planned administration of an influenza vaccine other than the study vaccines or of a vaccine not foreseen in the study protocol during the entire study period.
* Vaccination against influenza since January 2008 with a seasonal influenza vaccine.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the administration of the study vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of hypersensivity to a previous dose of influenza vaccine.
* History of allergy or reactions likely to be exacerbated by any component of the vaccine(s).
* Acute (active) clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by clinical evaluation (medical history and medical history directed physical examination) or pre-existing laboratory screening tests.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first administration of the study vaccine or planned administration during the study.
* Any medical conditions in which IM injections are contraindicated.
* Lactating female, female planning to become pregnant or planning to discontinue contraceptive precautions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2008-10-06; Primary Completion 2009-05-15 (Actual); Study Completion 2009-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (20):
- Germany (16):
  - GSK Investigational Site, Güglingen, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Rudersberg, Baden-Wurttemberg
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Rhaunen, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Freital, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Wolmirstedt, Saxony-Anhalt
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- GSK Investigational Site, Rotterdam, Netherlands
- Sweden (3):
  - GSK Investigational Site, Eskilstuna
  - GSK Investigational Site, Karlskrona
  - GSK Investigational Site, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 111737 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111737 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111737 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111737 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111737 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111737 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111737 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Started | 266 | 144 | 116
Completed | 261 | 142 | 111
Not Completed | 5 | 2 | 5
Not completed — Adverse Event | 5 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group | Total
Number analyzed (Participants) | 266 | 144 | 116 | 526
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.5 (5.27) | 73.8 (5.54) | 28.2 (6.34) | 63.59 (19.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 143 | 68 | 53 | 264
  Male | 123 | 76 | 63 | 262

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Adverse Events (AEs)
Description: Grade 3 ecchymosis, redness and swelling was greater than or equal to 100 millimeter (mm) i.e. ≥ 100 mm and grade 3 pain was considerable pain at rest, that prevented normal everyday activities. Any was occurrence of any local symptom regardless of their intensity grade.
Time Frame: Day 0-6
Population: The analysis was performed on Total Vaccinated cohort which included all subjects with the vaccine administration documented and symptom sheet completed.
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 265 | 144 | 115
Participants
  Any ecchymosis | 2 | 2 | 1
  Grade 3 ecchymosis | 0 | 0 | 0
  Any pain | 108 | 18 | 61
  Grade 3 pain | 0 | 0 | 0
  Any redness | 43 | 5 | 3
  Grade 3 redness | 1 | 0 | 0
  Any swelling | 20 | 7 | 1
  Grade 3 swelling | 0 | 0 | 0

2. Primary Outcome: Duration of Solicited Local AEs
Description: Duration was defined as number of days with any grade of local symptoms and grade for quantifiable symptoms: ecchymosis, redness and swelling was greater than (>) 20mm.
Time Frame: Day 0-6
Population: The analysis was performed on Total Vaccinated cohort which included all subjects with the vaccine administration documented and symptom sheet completed only on subjects that reported the specific symptom.
Measure: Median (Full Range); unit: Days
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 108 | 18 | 61
Days
  Ecchymosis: number analyzed (Participants) | 2 | 2 | 1
  Ecchymosis | 6.0 [6.0 to 6.0] | 4.0 [2.0 to 6.0] | 7.0 [7.0 to 7.0]
  Pain | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0] | 2.0 [1.0 to 7.0]
  Redness: number analyzed (Participants) | 43 | 5 | 3
  Redness | 2.0 [1.0 to 7.0] | 2.0 [2.0 to 3.0] | 2.0 [1.0 to 2.0]
  Swelling: number analyzed (Participants) | 20 | 7 | 1
  Swelling | 2.0 [1.0 to 7.0] | 3.0 [1.0 to 5.0] | 2.0 [2.0 to 2.0]

3. Primary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General AEs
Description: Any fever was defined as oral temperature ≥38.0 degree centigrade (°C), grade 3 fever was oral temperature >40.0°C. For other symptoms, any was defined as occurrence of any general symptom regardless of intensity grade or relationship to vaccination, grade 3 was defined as a general symptom that prevented normal activity and related was a general symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: Day 0-6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 265 | 144 | 115
Participants
  Any arthralgia | 30 | 6 | 10
  Grade 3 arthralgia | 0 | 0 | 0
  Related arthralgia | 20 | 5 | 7
  Any fatigue | 51 | 11 | 27
  Grade 3 fatigue | 1 | 0 | 2
  Related fatigue | 39 | 10 | 19
  Any gastrointestinal symptoms | 24 | 5 | 9
  Grade 3 gastrointestinal symptoms | 0 | 0 | 2
  Related gastrointestinal symptoms | 13 | 4 | 2
  Any headache | 39 | 7 | 30
  Grade 3 headache | 1 | 0 | 4
  Related headache | 24 | 4 | 17
  Any myalgia | 42 | 8 | 16
  Grade 3 myalgia | 0 | 0 | 0
  Related myalgia | 31 | 6 | 12
  Any shivering | 37 | 6 | 10
  Grade 3 shivering | 0 | 0 | 1
  Related shivering | 29 | 4 | 7
  Any fever | 5 | 1 | 5
  Grade 3 fever | 0 | 0 | 0
  Related fever | 4 | 1 | 3

4. Primary Outcome: Duration of Solicited General AEs
Description: Duration was defined as number of days with any grade of general symptoms.
Time Frame: Day 0-6
Population: as for outcome 2
Measure: Median (Full Range); unit: Days
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 51 | 11 | 30
Days
  Arthralgia: number analyzed (Participants) | 30 | 6 | 10
  Arthralgia | 2.0 [1.0 to 5.0] | 1.5 [1.0 to 3.0] | 3.0 [1.0 to 5.0]
  Fatigue: number analyzed (Participants) | 51 | 11 | 27
  Fatigue | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 5.0] | 2.0 [1.0 to 5.0]
  Gastrointestinal symptoms: number analyzed (Participants) | 24 | 5 | 9
  Gastrointestinal symptoms | 1.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0] | 1.0 [1.0 to 3.0]
  Headache: number analyzed (Participants) | 39 | 7 | 30
  Headache | 1.0 [1.0 to 7.0] | 1.0 [1.0 to 3.0] | 1.5 [1.0 to 4.0]
  Myalgia: number analyzed (Participants) | 42 | 8 | 16
  Myalgia | 2.0 [1.0 to 4.0] | 2.0 [2.0 to 5.0] | 2.0 [1.0 to 6.0]
  Shivering: number analyzed (Participants) | 37 | 6 | 10
  Shivering | 1.0 [1.0 to 6.0] | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Fever: number analyzed (Participants) | 5 | 1 | 5
  Fever | 1.0 [1.0 to 7.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]

5. Primary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited AEs
Description: Unsolicited adverse event (AE) covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade, grade 3 was unsolicited symptom that prevented normal activity and related was event assessed by the investigator as possibly related to the study vaccination.
Time Frame: Day 0-20
Population: The analysis was performed on Total Vaccinated cohort which included all subjects with the vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 266 | 144 | 116
Participants
  Any AE(s) | 49 | 20 | 18
  Grade 3 AE(s) | 6 | 1 | 4
  Related AE(s) | 1 | 2 | 0

6. Primary Outcome: Number of Subjects Reporting Any, Grade 3 and Related AEs With a Medically Attended Visit Between Day 0 to 20
Description: For each solicited and unsolicited AE the subject experienced, the subject was asked if they had received medical attention defined as hospitalization, an emergency room visit or a visit to or from medical personnel (medical doctor) for any reason. Any was defined as occurrence of any symptom regardless of intensity grade, grade 3 was defined as symptom that prevented normal activity and related was general symptom assessed by the investigator as possibly related to the study vaccination.
Time Frame: Day 0-20
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 266 | 144 | 116
Participants
  Any AE(s) | 20 | 8 | 9
  Grade 3 AE(s) | 4 | 1 | 1
  Related AE(s) | 0 | 0 | 0

7. Primary Outcome: Number of Subjects Reporting Any, Grade 3 and Related AEs With a Medically Attended Visit Between Day 21 to 179
Description: as for outcome 6
Time Frame: Day 21-179
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 266 | 144 | 116
Participants
  Any AE(s) | 103 | 48 | 33
  Grade 3 AE(s) | 26 | 8 | 9
  Related AE(s) | 0 | 0 | 0

8. Primary Outcome: Number of Subjects Reporting AEs of Specific Interest (AESI) Including Autoimmune Disease (AID)
Description: AESI for safety monitoring are a subset of AEs that include both clearly autoimmune diseases and also other inflammatory and/or neurologic disorders which may or may not have an autoiimune etiology. Any was defined as occurrence of any symptom regardless of intensity grade, grade 3 was defined as symptom that prevented normal activity and related was general symptom assessed by the investigator as possibly related to the study vaccination.
Time Frame: Day 0-179
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 266 | 144 | 116
Participants
  Any AE(s) | 0 | 0 | 0
  Grade 3 AE(s) | 0 | 0 | 0
  Related AE(s) | 0 | 0 | 0

9. Primary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs) Between Day 0 to Day 20
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade and related was event assessed by the investigator as causally related to the study vaccination.
Time Frame: Day 0-20
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 266 | 144 | 116
Participants
  Any SAE(s) | 4 | 2 | 1
  Related SAE(s) | 0 | 0 | 0

10. Primary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs) Between Day 21 to Day 179
Description: as for outcome 9
Time Frame: Day 21-179
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 266 | 144 | 116
Participants
  Any SAE(s) | 19 | 7 | 2
  Related SAE(s) | 0 | 0 | 0

11. Primary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs) From Day 180 to Day 209
Description: as for outcome 9
Time Frame: Day 180 to Day 209
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 266 | 144 | 116
Participants
  Any SAE(s) | 0 | 3 | 0
  Related SAE(s) | 0 | 0 | 0

12. Secondary Outcome: Haemagglutination Inhibition (HI) Antibody Titers at Days 0 and 21
Description: Antibody titers were expressed as Geometric mean titres (GMTs) with separate vaccine strains. The vaccine strains included A/Brisbane, A/Uruguay and B/Brisbane antigens.
Time Frame: At Day 0 and 21
Population: Analysis was performed on According-to-Protocol (ATP) immunogenicity cohort for HI which included all evaluable subjects for whom data concerning immunogenicity HI outcome measures were available at day 21.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 253 | 142 | 108
titer
  A/Brisbane vaccine strain at Day 0 | 27.9 [24.7 to 31.6] | 22.9 [19.6 to 26.7] | 43.2 [33.9 to 54.9]
  A/Brisbane vaccine strain at Day 21 | 74.6 [66.7 to 83.3] | 57.5 [49.5 to 66.8] | 164.7 [133.9 to 202.5]
  A/Uruguay vaccine strain at Day 0 | 28.1 [24.3 to 32.6] | 22.8 [19.0 to 27.4] | 28.9 [22.9 to 36.5]
  A/Uruguay vaccine strain at Day 21 | 243.9 [213.5 to 278.7] | 134.8 [107.9 to 168.4] | 171.1 [141.0 to 207.7]
  B/Brisbane vaccine strain at Day 0 | 126.5 [111.5 to 143.5] | 159.9 [136.1 to 188.0] | 192.7 [150.6 to 246.7]
  B/Brisbane vaccine strain at Day 21 | 519.0 [467.1 to 576.6] | 402.5 [344.2 to 470.6] | 711.5 [611.2 to 828.2]

13. Secondary Outcome: HI Antibody Titers at Day 180
Description: Antibody titers were expressed as GMTs with separate vaccine strains. The vaccine strains included A/Brisbane, A/Uruguay and B/Brisbane antigens.
Time Frame: Day 180
Population: Analysis was performed on According-to-Protocol (ATP) cohort for persistence which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available at day 180.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 241 | 130 | 103
titers
  A/Brisbane vaccine strain: number analyzed (Participants) | 240 | 130 | 103
  A/Brisbane vaccine strain | 34.9 [30.9 to 39.4] | 27.7 [23.9 to 32.0] | 99.5 [79.8 to 124.0]
  A/Uruguay vaccine strain: number analyzed (Participants) | 240 | 130 | 103
  A/Uruguay vaccine strain | 90.1 [77.0 to 105.4] | 69.9 [55.8 to 87.6] | 86.1 [68.2 to 108.7]
  B/Brisbane vaccine strain | 278.7 [248.4 to 312.6] | 255.7 [218.9 to 298.7] | 463.3 [384.0 to 558.9]

14. Secondary Outcome: The Number of Subjects Seropositive to HI Antibodies at Day 0 and 21
Description: Seropositivity was defined as antibody titer greater than or equal to the cut-off value i.e ≥ 1:10. The vaccine strains included A/Brisbane, A/Uruguay and B/Brisbane antigens.
Time Frame: At Day 0 and 21
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 253 | 142 | 108
Participants
  A/Brisbane vaccine strain at Day 0 | 226 | 125 | 97
  A/Brisbane vaccine strain at Day 21 | 251 | 141 | 108
  A/Uruguay vaccine strain at Day 0 | 212 | 116 | 90
  A/Uruguay vaccine strain at Day 21 | 253 | 140 | 108
  B/Brisbane vaccine strain at Day 0 | 253 | 142 | 108
  B/Brisbane vaccine strain at Day 21 | 253 | 142 | 108

15. Secondary Outcome: The Number of Subjects Seropositive to HI Antibodies at Day 180
Description: as for outcome 14
Time Frame: Day 180
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 241 | 130 | 103
Participants
  A/Brisbane vaccine strain: number analyzed (Participants) | 240 | 130 | 103
  A/Brisbane vaccine strain | 226 | 123 | 102
  A/Uruguay vaccine strain: number analyzed (Participants) | 240 | 130 | 103
  A/Uruguay vaccine strain | 235 | 125 | 99
  B/Brisbane vaccine strain | 241 | 130 | 103

16. Secondary Outcome: The Number of Subjects Seroconverted to HI Antibodies at Day 21
Description: Seroconversion was defined as the percentage of vaccinees who had either a pre-vaccination titre less than (<) 1:10 and a post-vaccination titre ≥1:40 or a pre-vaccination titre ≥1:10 and at least a 4-fold increase in post-vaccination titre. The vaccine strains included A/Brisbane, A/Uruguay and B/Brisbane antigens.
Time Frame: Day 21
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 253 | 142 | 108
Participants
  A/Brisbane vaccine strain | 77 | 46 | 48
  A/Uruguay vaccine strain | 209 | 97 | 67
  B/Brisbane vaccine strain | 130 | 47 | 50

17. Secondary Outcome: The Number of Subjects Seroconverted to HI Antibodies at Day 180
Description: Seroconversion was defined as the percentage of vaccinees who had either a pre-vaccination titre <1:10 and a post-vaccination titre ≥1:40 or a pre-vaccination titre ≥1:10 and at least a 4-fold increase in post-vaccination titre. The vaccine strains included A/Brisbane, A/Uruguay and B/Brisbane antigens.
Time Frame: Day 180
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 241 | 130 | 103
Participants
  A/Brisbane vaccine strain: number analyzed (Participants) | 240 | 130 | 103
  A/Brisbane vaccine strain | 15 | 11 | 31
  A/Uruguay vaccine strain: number analyzed (Participants) | 240 | 130 | 103
  A/Uruguay vaccine strain | 99 | 47 | 37
  B/Brisbane vaccine strain | 64 | 19 | 36

18. Secondary Outcome: HI Antibody Seroconversion Factor (SCF) at Day 21
Description: SCF was defined as the fold increase in serum HI GMTs post-vaccination compared to Day 0. The vaccine strains included A/Brisbane, A/Uruguay and B/Brisbane antigens.
Time Frame: Day 21
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: fold increase
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 253 | 142 | 108
fold increase
  A/Brisbane vaccine strain | 2.7 [2.4 to 3.0] | 2.5 [2.1 to 2.9] | 3.8 [3.0 to 4.9]
  A/Uruguay vaccine strain | 8.7 [7.5 to 9.9] | 5.9 [4.9 to 7.2] | 5.9 [4.8 to 7.3]
  B/Brisbane vaccine strain | 4.1 [3.6 to 4.6] | 2.5 [2.2 to 2.9] | 3.7 [3.0 to 4.5]

19. Secondary Outcome: HI Antibody SCF at Day 180
Description: as for outcome 18
Time Frame: Day 180
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: fold increase
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 241 | 130 | 103
fold increase
  A/Brisbane vaccine strain: number analyzed (Participants) | 240 | 130 | 103
  A/Brisbane vaccine strain | 1.3 [1.1 to 1.4] | 1.2 [1.1 to 1.4] | 2.4 [1.9 to 2.9]
  A/Uruguay vaccine strain: number analyzed (Participants) | 240 | 130 | 103
  A/Uruguay vaccine strain | 3.4 [3.0 to 3.8] | 2.9 [2.4 to 3.6] | 3.1 [2.5 to 3.9]
  B/Brisbane vaccine strain | 2.2 [2.0 to 2.4] | 1.7 [1.5 to 1.9] | 2.7 [2.3 to 3.2]

20. Secondary Outcome: The Number of Subjects Seroprotected to HI Antibodies at Day 0 and Day 21
Description: Seroprotection was defined as the percentage of vaccinees with a serum HI titre ≥1:40 that usually is accepted as indicating protection. The vaccine strains included A/Brisbane, A/Uruguay and B/Brisbane antigens.
Time Frame: At Day 0 and 21
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 253 | 142 | 108
Participants
  A/Brisbane vaccine strain at Day 0 | 124 | 55 | 68
  A/Brisbane vaccine strain at Day 21 | 222 | 108 | 101
  A/Uruguay vaccine strain at Day 0 | 121 | 58 | 53
  A/Uruguay vaccine strain at Day 21 | 248 | 123 | 104
  B/Brisbane vaccine strain at Day 0 | 236 | 136 | 101
  B/Brisbane vaccine strain at Day 21 | 253 | 141 | 108

21. Secondary Outcome: The Number of Subjects Seroprotected to HI Antibodies at Day 180
Description: as for outcome 20
Time Frame: Day 180
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 241 | 130 | 103
Participants
  A/Brisbane vaccine strain: number analyzed (Participants) | 240 | 130 | 103
  A/Brisbane vaccine strain | 143 | 65 | 89
  A/Uruguay vaccine strain: number analyzed (Participants) | 240 | 130 | 103
  A/Uruguay vaccine strain | 193 | 94 | 87
  B/Brisbane vaccine strain | 241 | 129 | 103

22. Secondary Outcome: The Geometric Mean (GM) Number of Influenza Specific Cluster of Differentiation 4 (CD4) T-cells Per Million CD4 T-cells for Each Vaccine Strain Expressing at Least Two Different Markers or Expressing Different Combinations of Markers at Days 0 and 21
Description: The markers assessed were CD4-ALL DOUBLES, CD40 Ligand (CD40L), interleukin 2 (IL-2), tumour necrosis factor alpha (TNF-α) and interferon gamma (IFN-γ) and vaccine strains tested included A/Brisbane, A/Uruguay and B/Brisbane antigens.
Time Frame: At Day 0 and 21
Population: Analysis was performed on According-to-Protocol (ATP) immunogenicity cohort for cell mediated immunity (CMI) which included subjects for whom data concerning immunogenicity CMI outcome measures were available at day 21.
Measure: Geometric Mean (Standard Deviation); unit: cells per million CD4 T-cells
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 66 | 34 | 22
cells per million CD4 T-cells
  A/Brisbane [CD4-ALL DOUBLES] Day 0 | 751.28 (492.55) | 682.47 (759.31) | 1179.17 (1031.92)
  A/Brisbane [CD4-ALL DOUBLES] Day 21: number analyzed (Participants) | 66 | 34 | 19
  A/Brisbane [CD4-ALL DOUBLES] Day 21 | 1431.41 (679.60) | 972.14 (1204.18) | 1513.30 (798.38)
  A/Uruguay [CD4-ALL DOUBLES] Day 0: number analyzed (Participants) | 65 | 33 | 22
  A/Uruguay [CD4-ALL DOUBLES] Day 0 | 451.86 (419.39) | 444.42 (578.82) | 743.45 (552.48)
  A/Uruguay [CD4-ALL DOUBLES] Day 21: number analyzed (Participants) | 66 | 32 | 19
  A/Uruguay [CD4-ALL DOUBLES] Day 21 | 912.85 (496.53) | 592.66 (518.19) | 912.28 (476.16)
  B/Brisbane [CD4-ALL DOUBLES] Day 0: number analyzed (Participants) | 65 | 34 | 22
  B/Brisbane [CD4-ALL DOUBLES] Day 0 | 828.74 (840.19) | 679.28 (702.37) | 1045.61 (510.95)
  B/Brisbane [CD4-ALL DOUBLES] Day 21: number analyzed (Participants) | 64 | 34 | 19
  B/Brisbane [CD4-ALL DOUBLES] Day 21 | 1361.30 (799.10) | 935.28 (1130.22) | 1403.64 (580.53)
  A/Brisbane [CD4-CD40L] Day 0 | 694.63 (452.67) | 616.27 (682.26) | 1127.82 (946.50)
  A/Brisbane [CD4-CD40L] Day 21: number analyzed (Participants) | 66 | 34 | 19
  A/Brisbane [CD4-CD40L] Day 21 | 1305.74 (622.93) | 855.81 (974.19) | 1379.47 (735.06)
  A/Uruguay [CD4-CD40L] Day 0: number analyzed (Participants) | 65 | 33 | 22
  A/Uruguay [CD4-CD40L] Day 0 | 392.35 (368.33) | 361.18 (498.91) | 646.92 (542.81)
  A/Uruguay [CD4-CD40L] Day 21: number analyzed (Participants) | 66 | 32 | 19
  A/Uruguay [CD4-CD40L] Day 21 | 803.34 (459.33) | 543.41 (463.96) | 816.08 (447.79)
  B/Brisbane [CD4-CD40L] Day 0: number analyzed (Participants) | 65 | 34 | 22
  B/Brisbane [CD4-CD40L] Day 0 | 775.18 (754.90) | 630.27 (630.81) | 959.42 (465.42)
  B/Brisbane [CD4-CD40L] Day 21: number analyzed (Participants) | 64 | 34 | 19
  B/Brisbane [CD4-CD40L] Day 21 | 1230.63 (731.08) | 850.96 (901.02) | 1275.70 (508.40)
  A/Brisbane [CD4-IFN-γ] Day 0 | 430.40 (373.24) | 338.29 (613.41) | 777.72 (837.25)
  A/Brisbane [CD4-IFN-γ] Day 21: number analyzed (Participants) | 66 | 34 | 19
  A/Brisbane [CD4-IFN-γ] Day 21 | 839.94 (536.38) | 481.04 (976.79) | 985.11 (713.98)
  A/Uruguay [CD4-IFN-γ] Day 0: number analyzed (Participants) | 65 | 33 | 22
  A/Uruguay [CD4-IFN-γ] Day 0 | 282.79 (321.42) | 301.64 (426.04) | 501.13 (482.16)
  A/Uruguay [CD4-IFN-γ] Day 21: number analyzed (Participants) | 66 | 32 | 19
  A/Uruguay [CD4-IFN-γ] Day 21 | 628.36 (400.49) | 399.84 (387.97) | 638.93 (418.36)
  B/Brisbane [CD4-IFN-γ] Day 0: number analyzed (Participants) | 65 | 34 | 22
  B/Brisbane [CD4-IFN-γ] Day 0 | 447.23 (708.32) | 299.25 (441.05) | 681.49 (413.65)
  B/Brisbane [CD4-IFN-γ] Day 21: number analyzed (Participants) | 64 | 34 | 19
  B/Brisbane [CD4-IFN-γ] Day 21 | 800.89 (648.91) | 478.15 (851.02) | 934.53 (471.32)
  A/Brisbane [CD4-IL2] Day 0 | 645.57 (445.17) | 542.90 (700.45) | 1033.28 (884.01)
  A/Brisbane [CD4-IL2] Day 21: number analyzed (Participants) | 66 | 34 | 19
  A/Brisbane [CD4-IL2] Day 21 | 1176.29 (568.05) | 816.63 (1114.87) | 1259.69 (691.36)
  A/Uruguay [CD4-IL2] Day 0: number analyzed (Participants) | 65 | 33 | 22
  A/Uruguay [CD4-IL2] Day 0 | 385.93 (375.33) | 392.63 (488.21) | 599.02 (523.72)
  A/Uruguay [CD4-IL2] Day 21: number analyzed (Participants) | 66 | 32 | 19
  A/Uruguay [CD4-IL2] Day 21 | 745.33 (428.75) | 505.78 (459.04) | 745.61 (444.27)
  B/Brisbane [CD4-IL2] Day 0: number analyzed (Participants) | 65 | 34 | 22
  B/Brisbane [CD4-IL2] Day 0 | 711.32 (760.06) | 547.71 (646.50) | 852.51 (479.69)
  B/Brisbane [CD4-IL2] Day 21: number analyzed (Participants) | 64 | 34 | 19
  B/Brisbane [CD4-IL2] Day 21 | 1112.52 (725.72) | 778.12 (1034.69) | 1156.73 (494.36)
  A/Brisbane [CD4-TNF-α] Day 0 | 606.82 (442.61) | 610.09 (669.96) | 900.67 (914.33)
  A/Brisbane [CD4-TNF-α] Day 21: number analyzed (Participants) | 66 | 34 | 19
  A/Brisbane [CD4-TNF-α] Day 21 | 1057.44 (568.35) | 749.70 (1068.11) | 1096.74 (689.90)
  A/Uruguay [CD4-TNF-α] Day 0: number analyzed (Participants) | 65 | 33 | 22
  A/Uruguay [CD4-TNF-α] Day 0 | 405.12 (403.06) | 414.27 (508.57) | 575.28 (509.48)
  A/Uruguay [CD4-TNF-α] Day 21: number analyzed (Participants) | 66 | 32 | 19
  A/Uruguay [CD4-TNF-α] Day 21 | 740.68 (448.67) | 449.51 (463.77) | 685.63 (429.55)
  B/Brisbane [CD4-TNF-α] Day 0: number analyzed (Participants) | 65 | 34 | 22
  B/Brisbane [CD4-TNF-α] Day 0 | 646.27 (718.92) | 558.87 (591.29) | 818.77 (441.82)
  B/Brisbane [CD4-TNF-α] Day 21: number analyzed (Participants) | 64 | 34 | 19
  B/Brisbane [CD4-TNF-α] Day 21 | 1021.43 (690.24) | 715.45 (973.99) | 1023.28 (475.97)

ADVERSE EVENTS:
Time Frame: Serious adverse events were assessed during Day 0-20, Day 21-179 and Day 180-209. Systematically assessed frequent adverse events (AEs) and non-systematically assessed frequent AEs were assessed during 7 and 21 day post vaccination period respectively.
Description: For the systematically assessed other (non-serious) adverse events, the number of participants at risk included those from Total Vaccinated Cohort who had the symptom sheet completed.
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Serious Adverse Events (participants affected / at risk) | 19/266 | 7/144 | 2/116
Other Adverse Events (participants affected / at risk) | 160/266 | 39/144 | 80/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | New Generation Influenza Vaccine GSK2186877A Group (N=266) | Fluarix Elderly Group (N=144) | Fluarix Young Group (N=116)
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 — SAE assessed from Day 0 to Day 20.
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 — SAE assessed from Day 0 to Day 20.
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 — SAE assessed from Day 0 to Day 20.
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 — SAE assessed from Day 0 to Day 20.
Locked-in syndrome (Nervous system disorders) | 1 | 0 | 0 — SAE assessed from Day 0 to Day 20.
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 — SAE assessed from Day 0 to Day 20.
Pneumonia (Infections and infestations) | 0 | 1 | 0 — SAE assessed from Day 0 to Day 20.
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 — SAE assessed from Day 0 to Day 20.
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 — SAE assessed from Day 0 to Day 20.
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 — SAE assessed from Day 0 to Day 20.
Testicular torsion (Reproductive system and breast disorders) | 0 | 0 | 1 — SAE assessed from Day 0 to Day 20.
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 — SAE assessed from Day 0 to Day 20.
Cerebrovascular accident (Nervous system disorders) | 3 | 0 | 0 — SAE assessed between Day 21 and Day 179.
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 — SAE assessed between Day 21 and Day 179.
Angina pectoris (Cardiac disorders) | 2 | 0 | 0 — SAE assessed between Day 21 and Day 179.
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0 — SAE assessed between Day 21 and Day 179.
Pneumonia (Infections and infestations) | 2 | 0 | 0 — SAE assessed between Day 21 and Day 179.
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 — SAE assessed between Day 21 and Day 179.
Anoxic encephalopathy (Nervous system disorders) | 0 | 1 | 0 — SAE assessed between Day 21 and Day 179.
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 — SAE assessed between Day 21 and Day 179.
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 — SAE assessed between Day 21 and Day 179.
Atrioventricular block (Cardiac disorders) | 1 | 0 | 0 — SAE assessed between Day 21 and Day 179.
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 — SAE assessed between Day 21 and Day 179.
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 — SAE assessed between Day 21 and Day 179.
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 — SAE assessed between Day 21 and Day 179.
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0 — SAE assessed between Day 21 and Day 179.
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 — SAE assessed between Day 21 and Day 179.
Convulsion (Nervous system disorders) | 0 | 1 | 0 — SAE assessed between Day 21 and Day 179.
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 — SAE assessed between Day 21 and Day 179.
Epididymitis (Reproductive system and breast disorders) | 1 | 0 | 0 — SAE assessed between Day 21 and Day 179.
Gastroenteritis norovirus (Infections and infestations) | 1 | 0 | 0 — SAE assessed between Day 21 and Day 179.
Glaucoma (Eye disorders) | 0 | 1 | 0 — SAE assessed between Day 21 and Day 179.
Hypertension (Vascular disorders) | 1 | 0 | 0 — SAE assessed between Day 21 and Day 179.
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 — SAE assessed between Day 21 and Day 179.
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0 — SAE assessed between Day 21 and Day 179.
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0 — SAE assessed between Day 21 and Day 179.
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 — SAE assessed between Day 21 and Day 179.
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 — SAE assessed between Day 21 and Day 179.
Sepsis (Infections and infestations) | 1 | 0 | 0 — SAE assessed between Day 21 and Day 179.
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0 — SAE assessed between Day 21 and Day 179.
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 — SAE assessed between Day 21 and Day 179.
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 — SAE assessed between Day 21 and Day 179.
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 — SAE assessed between Day 21 and Day 179.
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 — SAE assessed between Day 21 and Day 179.
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 — SAE assessed from Day 180.
Embolic cerebral infarction (Nervous system disorders) | 0 | 1 | 0 — SAE assessed from Day 180.
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 — SAE assessed from Day 180.
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 — SAE assessed from Day 180.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | New Generation Influenza Vaccine GSK2186877A Group (N=266) | Fluarix Elderly Group (N=144) | Fluarix Young Group (N=116)
Pain (General disorders) | 108/265 | 18 | 61/115
Redness (General disorders) | 43/265 | 5 | 3/115
Swelling (General disorders) | 20/265 | 7 | 1/115
Arthralgia (General disorders) | 30/265 | 6 | 10/115
Fatigue (General disorders) | 51/265 | 11 | 27/115
Gastrointestinal symptoms (General disorders) | 24/265 | 5 | 9/115
Headache (General disorders) | 39/265 | 7 | 30/115
Myalgia (General disorders) | 42/265 | 8 | 16/115
Shivering (General disorders) | 37/265 | 6 | 10/115
Nasopharyngitis (Infections and infestations) | 11 | 4 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.